CLINICAL TRIAL: NCT00350129
Title: Influence of Plasma Glucose Levels on Retinal Vascular Diameter and Choroidal Blood Flow in Vasospastic Subjects
Brief Title: Effect of Glucose on Ocular Blood Flow
Status: Completed | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Selim Orgul, University Hospital, Basel, Switzerland
Other Study IDs: 005-ZAC-2004-002
Record Dates: First submitted 2006-07-07; First posted 2006-07-10 (Estimated); Last update posted 2024-03-19 (Actual); Status verified 2024-03

CONDITIONS: Coronary Vasospasm
Keywords: glucose; vasospasm; RVA; LDF; vasospastic subjects; non-vasospastic subjects
MeSH Terms: conditions — Coronary Vasospasm

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: healthy vasospastic subjects
- 2: healthy non-vasospastic subjects

SUMMARY:
The primary objective is to assess the effect of glucose on retinal vascular diameter in otherwise healthy vasospastic subjects compared to non-vasospastic controls.

The secondary objective is to compare the effect of glucose also on choroidal blood flow in otherwise healthy vasospastic subjects with non-vasospastic controls.

DETAILED DESCRIPTION:
It is known that a glucose load can induce an increase in ocular blood flow. Acute hyperglycemia increases retinal vessel diameters in animals and humans. The purpose of this study is to compare the effect of glucose on the ocular blood flow in vasospastics and nonvasospastics. Body core temperature depends on basal metabolism. Peripheral vasoconstriction is a physiological way to preserve core temperature of the body. The etiology of primary vasospastic syndrome is unknown and potentially represents simply a reaction to a defective metabolism. Based on this hypothesis, vasospastics are expected to show a different vascular reaction to glucose.

On both study days, after an overnight fast, the subjects will be seated for 30 minutes in the Lab and local tropicamide will be applied for pupil dilatation. After stabilisation of blood pressure Retinal vessel diameter and choroidal blood flow will be assessed. Baseline blood glucose levels will be measured. Afterwards study substance (75 gram of Glucose or Aspartate) will be applied in 3 dl of water. One and a half hour later, the vascular measurements will be repeated. Ath the end of hemodynamic assessments, blood sugar level will be measured again.

ELIGIBILITY:
Inclusion Criteria:

* No history of the following problems: ocular or systemic disease; chronic or current systemic or topical medication; or of drug or alcohol abuse
* normal blood pressure (100-140 / 60-90 mmhg)
* best corrected visual acuity above 20/25 in both eyes
* no pathological findings upon a slit-lamp examination and indirect fundoscopy
* ametropia within -3 to +3 diopters of spherical equivalent
* less than 1 diopter astigmatism
* IOP < 20 mmHg in both eyes
* Subjects will be classified as vasospastic if they relate a clear history of frequent cold hands (answering yes to the questions: "do you have always cold hands, even during summer time?" and "do other people tell you that you have cold hands?") and as normals if they deny such a history
* Vasospastic propensity will also be assessed by capillaroscopy

Exclusion Criteria:

* Subjects describing "sometimes cold hands"
* if the test substance cannot be ingested
* not obtainable ocular blood flow measurements
* abnormally high levels of glucose at any point in time

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: healthy vasospastic subjects, healthy non-vasospastic subjects
Sampling Method: Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2002-12; Primary Completion 2003-02 (Actual); Study Completion 2003-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Selim Orgül, MD, Study Director — University Hospital, Basel, Switzerland
Locations (1):
- University Hospital Basel, Eye Clinic, Basel, Canton of Basel-City, Switzerland